CLINICAL TRIAL: NCT03724916
Title: A Phase 1b Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of TAK-079 in Combination With Standard Background Therapy in Patients With Moderate to Severe Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics (PK), and Pharmacodynamics (PD) of TAK-079 in Combination With Standard Background Therapy in Participants With Moderate to Severe Systemic Lupus Erythematosus (SLE)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-079-2001; U1111-1220-2497 (Other: World Health Organization)
Record Dates: First submitted 2018-10-18; First posted 2018-10-30 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-10

CONDITIONS: Systemic Lupus Erythematosus; Lupus Erythematosus, Systemic
Keywords: Drug therapy
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pooled Placebo (Placebo Comparator): TAK-079 placebo-matching injection, subcutaneously, once every 3 weeks in combination with principal investigator-directed background therapy for SLE for up to 12 weeks. Placebo data will be pooled across all the dose levels.
  Interventions: Drug: TAK-079 Placebo
- TAK-079 45 mg (Experimental): TAK-079 45 mg injection subcutaneously, once every 3 weeks in combination with principal investigator-directed background therapy for SLE for up to 12 weeks.
  Interventions: Drug: TAK-079
- TAK-079 90 mg (Experimental): TAK-079 90 mg injection subcutaneously, once every 3 weeks in combination with principal investigator-directed background therapy for SLE for up to 12 weeks.
  Interventions: Drug: TAK-079
- TAK-079 135 mg (Experimental): TAK-079 135 mg injection subcutaneously, once every 3 weeks in combination with principal investigator-directed background therapy for SLE for up to 12 weeks.
  Interventions: Drug: TAK-079

INTERVENTIONS:
Drug: TAK-079 — TAK-079 subcutaneous injection.
  Arms: TAK-079 135 mg; TAK-079 45 mg; TAK-079 90 mg
Drug: TAK-079 Placebo — TAK-079 placebo-matching subcutaneous injection.
  Arms: Pooled Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of TAK-079 in comparison with matching placebo, administered once every 3 weeks over a 12-week dosing period in participants with active SLE who are receiving stable background therapy for SLE.

DETAILED DESCRIPTION:
TAK-079 is being tested in a study population with moderate to severe SLE. This study will evaluate the safety and biologic activity of TAK-079 or matching placebo in combination with stable SLE background therapy.

The study will enroll approximately 24 participants across 3 sequentially enrolling cohorts. Each cohort will enroll 8 participants, where 6 participants will be assigned to TAK-079 injection, and 2 participants will be assigned to Placebo. Participants will receive TAK-079 or matching placebo in combination with principal investigator directed background therapy for SLE.

This multi-center trial will be conducted in the United States. Participants will make multiple visits to the clinic, and will be followed up for the safety assessment for the additional 12 weeks up to Week 24 after receiving their last dose of study drug. Based on the clinical assessments, participants may complete or may advance to long-term safety follow up period for an additional 12-week safety monitoring period up to Week 36.

ELIGIBILITY:
Inclusion Criteria:

1. The participant been diagnosed with SLE as defined by either the 2012 Systemic Lupus International Collaborating Clinics or the American College of Rheumatology diagnostic criteria.
2. The participant has a systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score greater than or equal to (>=) 6.
3. The participant is positive for anti-double-stranded deoxyribonucleic acid (dsDNA) antibodies and/or anti-extractable nuclear antigens (ENA) antibodies.

Exclusion Criteria:

1. The participant had an opportunistic infection less than or equal to (<=)12 weeks before initial study dosing or is currently undergoing treatment for a chronic opportunistic infection, such as tuberculosis (TB), pneumocystis pneumonia, cytomegalovirus, herpes simplex virus, herpes zoster, or atypical mycobacteria.
2. The participant currently has, or recently had, an acute or chronic infection requiring one or more of the following interventions: Hospitalization <=30 days before the screening visit. - Administered parenteral (IV or intramuscular) antibacterial, antiviral, antifungal, or antiparasitic agents <=30 days before the screening visit.
3. The participant has drug-induced SLE or any other rheumatologic or autoimmune disease (excluding secondary Sjögren syndrome or mixed connective tissue disease).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (19):
- United States (19):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - ACRC Studies, Poway, California
  - University of Colorado Denver, Aurora, Colorado
  - Clinical Research of West Florida - Clearwater, Clearwater, Florida
  - CRIA Research, Fort Lauderdale, Florida
  - Millennium Research, Ormond Beach, Florida
  - North Georgia Rheumatology Group-Duluth, Lawrenceville, Georgia
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Northwell Health, Great Neck, New York
  - State University of New York Upstate Medical Center (SUNY), Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Accurate Clinical Research, Houston, Texas
  - Southwest Rheumatology Research, LLC, Mesquite, Texas
  - Arthritis Northwest Rheumatology, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 13 investigative sites in United States from 26 November 2018 to 04 November 2021.
Pre-assignment Details: Participants with moderate to severe systemic lupus erythematosus (SLE) were sequentially enrolled to receive TAK-079 45 mg, TAK-079 90 mg, TAK-079 135 mg or TAK-079-matching placebo in a 3:1 ratio in this study.
Groups:
- Pooled Placebo: TAK-079 placebo-matching injection, subcutaneously, once every 3 weeks in combination with principal investigator-directed background therapy for SLE for up to 12 weeks. Placebo data was pooled across all the dose levels.
- TAK-079 45mg: TAK-079 45 mg injection subcutaneously, once every 3 weeks in combination with principal investigator-directed background therapy for SLE for up to 12 weeks.
Period: Overall Study
Arm/Group | Pooled Placebo | TAK-079 45mg | TAK-079 90 mg | TAK-079 135 mg
Started | 6 | 6 | 6 | 5
Safety Analysis Set (Safety analysis set included all participants who were enrolled and received at least 1 dose of study drug.) | 5 | 6 | 6 | 5
Pharmacokinetic (PK) Analysis Set (PK analysis set included all participants who received study drug and had at least 1 measurable serum concentration.) | 0 | 6 | 6 | 5
Pharmacodynamic (PD) Analysis Set (PD analysis set included all participants who received study drug and had at least 1 postdose PD measurement.) | 5 | 6 | 6 | 5
Immunogenicity Analysis Set (Immunogenicity analysis set consisted of all participants who received study drug and had a baseline and at least 1 postbaseline immunogenicity sample assessment.) | 5 | 6 | 5 | 5
Completed | 5 | 5 | 5 | 3
Not Completed | 1 | 1 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 2
Not completed — Randomized but not Treated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | TAK-079 45mg | TAK-079 90 mg | TAK-079 135 mg | Total
Number analyzed (Participants) | 5 | 6 | 6 | 5 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (6.58) | 51.0 (22.01) | 46.7 (6.53) | 49.6 (13.50) | 46.2 (14.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 4 | 20
  Male | 0 | 0 | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 1 | 4
  Not Hispanic or Latino | 4 | 4 | 6 | 4 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 1 | 2 | 9
  White | 3 | 2 | 4 | 1 | 10
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Treatment-emergent Adverse Event (TEAE) and Serious Adverse Event (SAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an AE with an onset that occurs after receiving study drug. An SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From the study start to end of the study (up to Week 36)
Population: Safety analysis set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | TAK-079 45mg | TAK-079 90 mg | TAK-079 135 mg
Number analyzed (Participants) | 5 | 6 | 6 | 5
Participants
  TEAEs | 3 | 4 | 6 | 2
  SAEs | 0 | 1 | 0 | 1

2. Primary Outcome: Number of Participants With Grade 3 or Higher Treatment Emergent Adverse Events (TEAEs)
Description: The severity of TEAEs will be graded using National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.0 definitions of Grade 1 through Grade 5. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: From the study start up to end of the study (up to Week 36)
Population: Safety analysis set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | TAK-079 45mg | TAK-079 90 mg | TAK-079 135 mg
Number analyzed (Participants) | 5 | 6 | 6 | 5
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With ≥ 1 Adverse Event (AE) Leading to Treatment Discontinuation
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug.
Time Frame: From the study start up to end of the study (up to Week 36)
Population: Safety analysis set consisted of all participants who were enrolled and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | TAK-079 45mg | TAK-079 90 mg | TAK-079 135 mg
Number analyzed (Participants) | 5 | 6 | 6 | 5
Participants | 0 | 0 | 0 | 1

4. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for TAK-079
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose; Day 22 pre-dose and at multiple time points (up to 108 hours) post-dose; Days 43 and 64 pre-dose and at multiple time points (up to 5 hours) post-dose
Population: Pharmacokinetics analysis set consisted of all participants who received study drug and had at least 1 measurable serum concentration. Number analyzed is the number of participants available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | TAK-079 45mg | TAK-079 90 mg | TAK-079 135 mg
Number analyzed (Participants) | 6 | 6 | 5
nanograms per millilitre (ng/mL)
  Day 1 | 57.5 (71.7) | 660.0 (1050) | 6130 (5170)
  Day 22: number analyzed (Participants) | 6 | 5 | 5
  Day 22 | 95.4 (187) | 1570 (2930) | 6330 (9450)
  Day 43: number analyzed (Participants) | 6 | 4 | 4
  Day 43 | 10.6 (17.5) | 1440 (2550) | 559 (714)
  Day 64: number analyzed (Participants) | 6 | 4 | 4
  Day 64 | 16.4 (17.4) | 568 (841) | 3100 (3900)

5. Secondary Outcome: AUClast: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for TAK-079
Time Frame: as for outcome 4
Population: As pre-specified in SAP, data for AUClast was not evaluated due to sparse PK sampling.
Arm/Group | Pooled Placebo | TAK-079 45mg | TAK-079 90 mg | TAK-079 135 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Change From Baseline In Immune Cell Subsets
Description: Immune cell subsets included plasma cells, plasma blast (PBs), natural killer (NK) cells, B cells, T cells, monocytes, and total lymphocytes. The concentration of each plasma subset cell type is measured at baseline and post-baseline timepoints and the number of participants who had change in the concentration of each plasma subset cells from baseline were evaluated and reported in this outcome measure.
Time Frame: Baseline up to Day 85 (End of Treatment [EOT])
Population: PD analysis set included all participants who received study drug and had at least 1 postdose PD measurement. Overall number analyzed are the number of participants who had baseline and post-baseline data for change.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | TAK-079 45mg | TAK-079 90 mg | TAK-079 135 mg
Number analyzed (Participants) | 4 | 6 | 4 | 4
Participants
  Participants who had change in Plasma cell concentration | 4 | 6 | 4 | 4
  Participants who had change in Plasmablasts concentration | 4 | 6 | 4 | 4
  Participants who had change in NK cells concentration | 4 | 6 | 4 | 4
  Participants who had change in B cells concentration | 4 | 6 | 4 | 4
  Participants who had change in T cells concentration | 4 | 6 | 4 | 4
  Participants who had change in Monocytes concentration | 4 | 6 | 4 | 4
  Participants who had change in Lymphocytes concentration | 4 | 6 | 4 | 4

7. Secondary Outcome: Number of Participants With Change From Baseline in Immune Cell Subsets Determined Based on Receptor Occupancy
Description: Receptor occupancy was evaluated for plasma cells, PBs, NK cells, B cells, T cells, and monocytes. The concentration of cells expressing CD38+ and those not expressing the same is correlated and used to determine receptor occupancy. The receptor occupancy of these cells was determined at baseline and post-baseline timepoints. The number of participants who had change in the receptor occupancy of these cells from baseline were evaluated and reported in this outcome measure.
Time Frame: Baseline up to Day 85 (EOT)
Population: Pharmacokinetics analysis set consisted of all participants who received study drug and had at least 1 measurable serum concentration. Overall number analyzed are the number of participants who had baseline and post-baseline data.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | TAK-079 45mg | TAK-079 90 mg | TAK-079 135 mg
Number analyzed (Participants) | 4 | 6 | 4 | 4
Participants
  Participants who had change in receptor occupancy: Plasma Cells | 4 | 3 | 4 | 4
  Participants who had change in receptor occupancy: Plasmablasts | 4 | 5 | 4 | 4
  Participants who had change in receptor occupancy: CD38+NK cells | 4 | 5 | 4 | 4
  Participants who had change in receptor occupancy: CD38+B cells | 4 | 5 | 4 | 4
  Participants who had change in receptor occupancy: CD38+T cells | 4 | 5 | 4 | 4
  Participants who had change in receptor occupancy: CD38+Monocytes | 4 | 5 | 4 | 4

8. Secondary Outcome: Change From Baseline in Cytokines Level
Time Frame: Baseline up to Day 85
Population: Since no participants had potential symptoms of cytokine release syndrome (CRS) or developed a CRS while on study, the assessment for cytokines was never performed.
Arm/Group | Pooled Placebo | TAK-079 45mg | TAK-079 90 mg | TAK-079 135 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies
Time Frame: Baseline up to Day 85 (EOT)
Population: Immunogenicity set consisted of all participants who received study drug and had a baseline and at least 1 postbaseline immunogenicity sample assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Placebo | TAK-079 45mg | TAK-079 90 mg | TAK-079 135 mg
Number analyzed (Participants) | 5 | 6 | 5 | 5
Participants
  Baseline | 3 | 0 | 1 | 1
  EOT | 3 | 2 | 0 | 2

ADVERSE EVENTS:
Time Frame: From the study start up to end of the study (up to Week 36)
Description: Safety analysis set included all subjects who were enrolled and received at least 1 dose of study drug.
Arm/Group | Pooled Placebo | TAK-079 45mg | TAK-079 90 mg | TAK-079 135 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/6 | 0/6 | 1/5
Other Adverse Events (participants affected / at risk) | 3/5 | 4/6 | 6/6 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=5) | TAK-079 45mg (N=6) | TAK-079 90 mg (N=6) | TAK-079 135 mg (N=5)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=5) | TAK-079 45mg (N=6) | TAK-079 90 mg (N=6) | TAK-079 135 mg (N=5)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Bezoar (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestinal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2019-03-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT03724916/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT03724916/SAP_001.pdf